CLINICAL TRIAL: NCT04675125
Title: A Prospective Study of Application of Platelet Mapping in Chronic Liver Disease Complicated With ALI and/or AD in China
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2020-052
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-07

CONDITIONS: Thrombelastography, Acute Liver Injury, Acute Decompensation, Platelet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ineffective hemostasis or a paradoxical prothrombotic state of Acute-on-chronic liver disease (ACLF) has been well established. Thrombelastography measures the dynamics of thrombin production and provides a global assessment of coagulation incorporating the cumulative effect of the interactions at various levels between plasma components and cellular component of coagulation. Through the previous studies(NCT03281278 and NCT04119973), we found that ACLF patients with high ADP inhibition rate had high 28-day mortality.This study aims to validate that high ADP inhibition rate only occurs in patients with liver failure and is related to the severity of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. chronic liver disease: including chronic liver hepatitis patients without cirrhosis, compensated cirrhosis patients, decompensated cirrhosis patients and non-alcoholic fatty liver disease patients.
2. ALI(acute liver injury): including [ALT > 3 ULN(upper limited of normal),AST > 3 ULN or TB > 2 ULN within 1 week before enrollment] or AD(acute decompensation) : including [(having ascites, hepatic encephalopathy and/or bacterial infection within 1 month before enrollment)].

Exclusion Criteria:

1. those who had hepatocellular carcinoma or other types of malignancies;
2. obstructive biliary diseases or other disease lead to bilirubin evaluation;
3. those who had acute hemorrhage one week before admission
4. those who received platelet, cryo transfusion or plasmapheresis one week before admission
5. pregnancy and breastfeeding
6. those who received liver transplantation or kidney transplantation;
7. combine with other disease lead to organ failure including heart failure (NYHA IV),respiratory failure（PaO2<60mmHg),renal insufficiency(CKD 5) and conscious disturbance (GCS<8)
8. readmission;
9. death within 24 hours.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic liver disease patients（with liver dysfunction more than 6 months） with acute liver injury[with ALT>3 ULN),AST>3NL or TB>2 ULN within 1 week before enrollment] or acute decompensation[having ascites, hepatic encephalopathy and/or bacterial infection within 1 month before enrollment].
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-05 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28-day
  death within 28-day

SECONDARY OUTCOMES:
28-day progression | 28-day
  progressed to EASL defined ACLF
90-day mortality | 90-day
  death within 90-day

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China